CLINICAL TRIAL: NCT07322861
Title: A Controlled Trial Comparing Virtual Reality-Based PABLO Training With Traditional Otago Physiotherapy for Balance, Frailty, and Fall Risk in Adults Aged 45 Years and Older
Brief Title: Virtual Reality-Based vs Traditional Physiotherapy for Balance, Frailty, and Fall Prevention in Adults Aged 45 Years and Older
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Dr. Hammad Alhasan, Dr, Umm Al-Qura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAPO-02-K-012-2025-11-2975
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Falls; Balance Deficits; Mobility Limitations
Keywords: Virtual Reality Rehabilitation; Balance Training; Fall Prevention; Frailty; Exergaming
MeSH Terms: conditions — Frailty; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: This is a 12-week, two-arm, parallel-group interventional study comparing VR-based PABLO training with traditional Otago-based physiotherapy. Participants attend supervised sessions twice weekly (30 minutes each), with outcomes assessed at baseline (week 0) and post-intervention (week 12).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to group allocation. Participants and treating physiotherapists are not blinded due to the nature of the interventions. Data analysts will receive de-identified datasets labeled by group codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-Based Training Program (Experimental)
  Interventions: Device: Virtual Reality-Based Training Program
- Traditional Physiotherapy Program (Active Comparator)
  Interventions: Other: Physiotherapy Exercise Program

INTERVENTIONS:
Device: Virtual Reality-Based Training Program — Participants assigned to this arm will receive a virtual reality (VR)-based exercise program using the PABLO system. The intervention will be delivered over 12 weeks, with two supervised sessions per week (approximately 30 minutes per session). Training will include interactive balance exercises with real-time biofeedback, strength and power tasks, aerobic stepping activities, and flexibility exercises. Exercise intensity and progression will be guided by perceived exertion and task performance. The program is designed to improve balance control, mobility, strength, and engagement while reducing fall risk
  Arms: Virtual Reality-Based Training Program
Other: Physiotherapy Exercise Program — Participants assigned to this arm will receive a traditional physiotherapy program based on the Otago Exercise Programme. The intervention will be delivered over 12 weeks, with two supervised sessions per week (approximately 30 minutes per session). The program will include balance training, lower-limb strength and power exercises, aerobic components, and flexibility exercises, following established Otago progression principles. This program aims to improve balance, mobility, and physical function and reduce fall risk using conventional physiotherapy methods.
  Arms: Traditional Physiotherapy Program

SUMMARY:
This study will compare two exercise-based rehabilitation programs to improve balance and reduce fall risk in adults aged 45 years and older who have had at least one fall in the past year or have balance problems. Participants will be assigned to one of two groups: (1) a virtual reality (VR) exercise program using the PABLO system, or (2) a traditional physiotherapy program based on the Otago approach. Both programs will include balance training, strength/power exercises, aerobic activity, and flexibility. The program will last 12 weeks, with two supervised sessions per week (about 30 minutes each). Assessments will be completed at the start of the study and again after 12 weeks. The main outcomes include frailty status, number of falls, mobility (Timed Up and Go test), and balance (Berg Balance Scale). Additional outcomes include grip strength, quality of life (SF-12), and program adherence and safety. The study will help determine whether VR-based rehabilitation improves participation and outcomes compared with traditional physiotherapy.

DETAILED DESCRIPTION:
Falls and frailty are major contributors to functional decline, loss of independence, and reduced quality of life in middle-aged and older adults. Balance impairment, muscle weakness, and fear of falling often coexist and interact, creating a cycle of reduced physical activity, deconditioning, and increased fall risk. Exercise-based physiotherapy programs, such as the Otago program, are effective for fall prevention; however, long-term adherence remains a major challenge, particularly in unsupervised or home-based settings. Poor adherence can substantially limit the clinical benefits of rehabilitation.

Virtual reality (VR)-based rehabilitation has emerged as a promising approach to address these challenges by improving engagement, motivation, and task-specific motor learning through real-time feedback and interactive exercises. Sensor-based VR systems, such as the PABLO system, allow targeted training of balance, strength, and functional movements while providing objective performance feedback. Although VR interventions have shown beneficial effects on balance and mobility in older adults, direct comparisons with conventional physiotherapy programs in adults at risk of falls remain limited.

This study is designed to compare the effects of a VR-based PABLO training program with a traditional Otago-based physiotherapy program in adults aged 45 years and older who have a history of falls or balance dysfunction. Participants will undergo a 12-week intervention consisting of twice-weekly, supervised exercise sessions. Both programs are structured to include balance training, strength and power exercises, aerobic components, and flexibility, with balance and strength emphasized as core elements.

The study will evaluate changes in frailty status, fall frequency, balance, mobility, grip strength, and quality of life from baseline to post-intervention. In addition, adherence, compliance, and safety outcomes will be monitored to assess feasibility and tolerability of both approaches. By comparing a technology-enhanced rehabilitation program with a well-established traditional physiotherapy model, this trial aims to generate evidence to inform clinical decision-making and support the integration of VR-based interventions into fall prevention and frailty management strategies for adults at increased risk of functional decline.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 40 years and older
* History of at least one fall in the past 12 months OR clinical evidence of balance dysfunction
* Ability to walk at least 10 meters, with or without an assistive device
* Adequate cognitive function, defined as Mini-Mental State Examination (MMSE) score ≥ 24
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Severe cognitive impairment (MMSE < 24)
* Unstable cardiovascular, musculoskeletal, or neurological conditions that contraindicate exercise participation
* Severe uncorrected visual or auditory impairment that interferes with training or assessments
* Current participation in another structured exercise or rehabilitation program
* Any medical condition deemed unsafe for participation by the treating physiotherapist

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Frailty Status (Arabic FRAIL Scale) | Baseline (Week 0) and Post-Intervention (Week 12)
  Frailty will be assessed using the validated Arabic FRAIL scale, which includes five domains: fatigue, resistance, ambulation, illnesses, and weight loss. Scores range from 0 (robust) to 5 (frail), with higher scores indicating greater frailty.
Balance Performance (Berg Balance Scale) | Baseline (Week 0) and Post-Intervention (Week 12)
  Balance will be measured using the Berg Balance Scale (BBS), a 14-item clinical test of static and dynamic balance. Total scores range from 0 to 56, with lower scores indicating poorer balance and higher fall risk.
Functional Mobility (Timed Up and Go Test) | Time Frame: Baseline (Week 0) and Post-Intervention (Week 12)
  Functional mobility will be assessed using the Timed Up and Go (TUG) test, which measures the time (in seconds) required to stand up from a chair, walk 3 meters, turn, return, and sit down. Longer times indicate greater mobility impairment and increased fall risk.

SECONDARY OUTCOMES:
Number of Falls | Baseline (previous 12 months) and During Intervention (Weeks 1-12)
  Falls will be recorded using retrospective 12-month fall history at baseline and a prospective falls diary during the intervention period.
Grip Strength | Baseline (previous 12 months) and During Intervention (Weeks 1-12)
  Handgrip strength measured using a Jamar dynamometer or PABLO hand sensors. Three trials will be performed on the dominant hand, with the best value (kg) recorded.
Quality of Life (SF-12) | Baseline (previous 12 months) and During Intervention (Weeks 1-12)
  Health-related quality of life assessed using the SF-12 questionnaire, covering physical and mental health domains.

OTHER OUTCOMES:
Age | Baseline (Week 0)
  Age in years
Weight | Baseline (Week 0)
  Weight in kilograms
Height | Baseline (Week 0)
  height in centimetre
Body mass index | Baseline (Week 0)
  weight and height will be combined to report BMI in kg/m^2
Number of Morbidities | Baseline (Week 0)
  The number of chronic medical conditions will be recorded for each participant based on self-report at baseline. Conditions will be summed to generate a total morbidity count, with higher values indicating greater multimorbidity burden.
Presence of Musculoskeletal Pain | Baseline (Week 0)
  The presence of musculoskeletal pain will be recorded based on participant self-report. Pain will be classified as present or absent at the time of assessment.
Smoking Status | Baseline (Week 0)
  Smoking status will be recorded based on participant self-report and classified as current smoker or non-smoker at baseline.
Specific chronic diseases | Baseline (Week 0)
  The presence of specific chronic diseases will be recorded at baseline based on participant self-report. Conditions assessed will include physician-diagnosed hypertension, diabetes mellitus, cardiovascular disease, and other chronic conditions. Each condition will be recorded as present or absent.
Polypharmacy Status | Baseline (Week 0)
  Polypharmacy will be assessed at baseline based on participant self-report of regular medication use. Polypharmacy will be defined as the concurrent use of five or more medications and recorded as present or absent.
Intervention Adherence | Throughout Intervention (Weeks 1-12)
  Adherence assessed as the percentage of attended sessions out of the planned 24 sessions and completion of prescribed exercises or VR tasks.
Safety and Adverse Events | Throughout Intervention (Weeks 1-12)
  * Falls occurring during supervised intervention sessions will be recorded using a standardized adverse event log.
  * Episodes of dizziness reported or observed during intervention sessions will be recorded as adverse events.
  * New or worsened musculoskeletal pain occurring during or immediately after intervention sessions will be recorded as adverse events.
  * Cardiovascular symptoms, including chest discomfort, palpitations, shortness of breath, or abnormal cardiovascular responses during training sessions, will be recorded as adverse events.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to ethical and confidentiality considerations. The informed consent obtained from participants does not include permission for public sharing of de-identified individual-level data. Aggregate study results will be reported through publications and presentations.